CLINICAL TRIAL: NCT00355303
Title: Comparison of Misoprostol and PGE2 Gel for Induction of Labour in in Premature Rupture of Membranes at Term- A Randomized Comparative Trial
Brief Title: Comparison of Misoprostol and Prostaglandin E2 (PGE2) Gel for Induction of Labour in Premature Rupture of Membranes at Term
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nilratan Sircar Medical College (Other Government)
Responsible Party: Principal Investigator, Dr Snehamay Chaudhuri, Associate Professor , Obstetrics and Gynecology, NRS Medical College, Nilratan Sircar Medical College
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2-Chaudhuri
Record Dates: First submitted 2006-07-19; First posted 2006-07-21 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Premature Rupture of Membranes at Term
Keywords: Premature rupture of membranes at term; Induction of labour; Misoprostol; PGE2 gel; Immediate induction with PGE2 gel; Immediate induction with Misoprostol
MeSH Terms: interventions — Misoprostol; Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Misoprostol tablet, PGE2 gel (Active Comparator): participants are assigned to one of two arms for the duration of the study In one group induction of labour is done by intravaginal misoprostol tablets at 4 hrly interval with maximum of five doses.In other group PGE2 gel is applied in poaterior fornix at six hourly interval.
  Interventions: Drug: Misoprostol; Drug: PGE2 gel

INTERVENTIONS:
Drug: Misoprostol — Vaginal application of Misoprostol tablets at 4 hrly interval with maximumof five doses
  Other Names: Misoprost
Drug: PGE2 gel — PGE2 gel will be applied in poaterior fornix at six hrly interval with maximum of 2 doses
  Other Names: Dinoprostone gel

SUMMARY:
The purpose of this study is to determine whether induction of labor with vaginal misoprostol application will result in fewer cesarean deliveries than vaginal PGE2 gel application in women with premature rupture of membranes at term.

ELIGIBILITY:
Inclusion Criteria:

* Premature rupture of membranes at 37 or more weeks
* Single live fetus in cephalic presentation

Exclusion Criteria:

* Women in labour
* Women with contraindication of induction of labour
* Women with previous caesarean section or uterine surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 932 (Actual)
Dates: Start 2006-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Caesarean Section rate | 48 hours

SECONDARY OUTCOMES:
Induction delivery time | 48 hours
Neonatal & maternal infectious morbidity | 14 days following date of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Snehamay Chaudhuri, MBBS,MD.DNB, Principal Investigator — Nilratan Sircar Medical College , Kolkata, West bengal , India
Locations (1):
- Nilratan Sircar Medical College, 138,AJC Bose Road,, Kolkata, West Bengal, India